CLINICAL TRIAL: NCT05775757
Title: Registry for Analysis of Impact of Radiation Dose to Skin on Cosmetic Outcome and Patient-reported Outcomes in Patients With Breast Cancer Treated With Radiation Therapy
Brief Title: SMC Radiation Oncology Breast Cancer Cohort Study
Acronym: RASCO
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Haeyoung Kim, Associate professor, Samsung Medical Center
Other Study IDs: SMC 2021-05-045
Record Dates: First submitted 2023-02-15; First posted 2023-03-20 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Radiotherapy Side Effect
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Hypofractionated radiation therapy — Both 3-week and 1-week hypofractioanted radiation therapy are allowed. (simultaneous or sequential tumor bed boost is allowed.) A 3-week regimen includes 42.4 Gy in 16 fractions. A 1-week regimen includes 26 Gy in 5 fractions or 28.5 Gy in 3 fractions, 30 Gy in 5 fractions.

SUMMARY:
The goal of this observational study is to learn about toxicities and cosmetic outcomes in breast cancer patients treated with hypofractionated radiotherapy.

The main question it aims to answer are:

* Changes in breast skin
* Factors related to breast skin changes
* Patient-reported outcomes
* Cosmetic outcomes

Participants will be assessed by multi-dimensional methods before and after radiotherapy:

* Photographs
* Fibrometer
* Questionnaires (BREAST-Q)
* CTCAE version 4.03 evaluated by treating physicians

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer treated with curative surgery

Exclusion Criteria:

* History of thoracic radiation therapy

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Any breast cancer patients treated with curative surgery is eligible except for history of thoracic radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of cosmesis from baseline | After 2-3 weeks after the start of radiation therapy (During radiation therapy)
  Evaluated by two blinded independent physicians based on photographs
Change of cosmesis from baseline | 2-3 weeks after the completion of radiation therapy
  Evaluated by two blinded independent physicians based on photographs
Change of cosmesis from baseline | 6 months after radiation therapy
  Evaluated by two blinded independent physicians based on photographs
Change of cosmesis from baseline | 1 year after radiation therapy
  Evaluated by two blinded independent physicians based on photographs
Change of cosmesis from baseline | 2 year after radiation therapy
  Evaluated by two blinded independent physicians based on photographs
Change of cosmesis from baseline | 5 year after radiation therapy
  Evaluated by two blinded independent physicians based on photographs
Change of fibrosis from baseline | After 2-3 weeks after the start of radiation therapy (During radiation therapy)
  Evaluated using fibrometer measuring both breast
Change of fibrosis from baseline | 2-3 weeks after the completion of radiation therapy
  Evaluated using fibrometer measuring both breast
Change of fibrosis from baseline | 6 months after radiation therapy
  Evaluated using fibrometer measuring both breast
Change of fibrosis from baseline | 1 year after radiation therapy
  Evaluated using fibrometer measuring both breast
Change of fibrosis from baseline | 2 year after radiation therapy
  Evaluated using fibrometer measuring both breast
Change of fibrosis from baseline | 5 year after radiation therapy
  Evaluated using fibrometer measuring both breast
Change of patient-reported outcome from baseline | After 2-3 weeks after the start of radiation therapy (During radiation therapy)
  BREAST-Q questionnaire is used to evaluate patient-reported outcome.
Change of patient-reported outcome from baseline | 2-3 weeks after the completion of radiation therapy
  BREAST-Q questionnaire is used to evaluate patient-reported outcome.
Change of patient-reported outcome from baseline | 6 months after radiation therapy
  BREAST-Q questionnaire is used to evaluate patient-reported outcome.
Change of patient-reported outcome from baseline | 1 year after radiation therapy
  BREAST-Q questionnaire is used to evaluate patient-reported outcome.
Change of patient-reported outcome from baseline | 2 year after radiation therapy
  BREAST-Q questionnaire is used to evaluate patient-reported outcome.
Change of patient-reported outcome from baseline | 5 year after radiation therapy
  BREAST-Q questionnaire is used to evaluate patient-reported outcome.
Physician assessed toxicity | After 2-3 weeks after the start of radiation therapy
  CTCAE version 4.03 is used to evaluate physician-assessed toxicities.
Physician assessed toxicity | 2-3 weeks after the completion of radiation therapy
  CTCAE version 4.03 is used to evaluate physician-assessed toxicities.
Physician assessed toxicity | 6 months after radiation therapy
  CTCAE version 4.03 is used to evaluate physician-assessed toxicities.
Physician assessed toxicity | 1 year after radiation therapy
  CTCAE version 4.03 is used to evaluate physician-assessed toxicities.
Physician assessed toxicity | 2 year after radiation therapy
  CTCAE version 4.03 is used to evaluate physician-assessed toxicities.
Physician assessed toxicity | 5 year after radiation therapy
  CTCAE version 4.03 is used to evaluate physician-assessed toxicities.

CONTACTS AND LOCATIONS:
Overall Officials: Haeyoung Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No